CLINICAL TRIAL: NCT03783416
Title: Safety of Ixazomib Targeting Plasma Cells in Multiple Sclerosis: A Phase 1b Randomised, Double-blind, Placebo-controlled Trial.
Brief Title: SIZOMUS Safety of Ixazomib Targeting Plasma Cells in Multiple Sclerosis
Acronym: SIZOMUS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Queen Mary University of London (Other)
Collaborators: Takeda Pharmaceuticals International, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 012436; 2018-003686-34 (EudraCT Number)
Record Dates: First submitted 2018-12-10; First posted 2018-12-21 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Relapsing Remitting Multiple Sclerosis; Primary Progressive Multiple Sclerosis; Secondary Progressive Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive | interventions — ixazomib; Capsules

STUDY DESIGN:
Intervention Model Description: This is a double-blind, randomised, placebo-controlled trial. Randomisation will be stratified by disease stage, i.e. RRMS (and established on DMT) versus progressive MS (and not on DMT). The expected study duration is 36 months (a 12-month recruitment period and a 24-month treatment period). There will be 72 participants: 48 on ixazomib; 24 on placebo.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ixazomib (NINLARO®) (Experimental): Treatment will follow a 28-day cycle. Participants will take one Ixazomib (NINLARO) capsule orally on days 1, 8, and 15 of each 28-day cycle, followed by one treatment-free week, in sequence, for the duration of the trial.
  Interventions: Drug: Ixazomib (NINLARO®) capsules / Matching placebo capsules
- Placebo (Placebo Comparator): Treatment will follow a 28-day cycle. Participants will take one placebo capsule orally on days 1, 8, and 15 of each 28-day cycle, followed by one treatment-free, in sequence, for the duration of the trial.
  Interventions: Drug: Ixazomib (NINLARO®) capsules / Matching placebo capsules

INTERVENTIONS:
Drug: Ixazomib (NINLARO®) capsules / Matching placebo capsules — Participants will be treated for a maximum of 24 months

SUMMARY:
The study seeks to investigate safety and efficacy of ixazomib (NINLARO), a proteasome inhibitor, in multiple sclerosis (MS). Participants will receive either ixazomib capsules or placebo capsules for up to 24 months.

DETAILED DESCRIPTION:
The production of antibodies in the form of oligoclonal bands (OCBs) from plasma cells (cells involved in the body's immune response), is the hallmark of MS. Recent evidence suggests that plasma cells are resident in the meninges (protective membranes of the brain and spinal cord) of people with Multiple Sclerosis (pwMS). Ixazomib is a drug which has been effective in treating multiple myeloma, a disease caused by aberrant plasma cells. The purpose of this study is to investigate whether ixazomib can reduce or clear OCBs from the cerebrospinal fluid (CSF) of pwMS. Participants will be randomly assigned to receive either ixazomib capsules (active drug arm) or placebo capsules (placebo arm) for up to 24 months. Participants with relapsing remitting MS (who are stable on disease modifying therapy) and those with progressive MS (who are not on disease modifying therapy) will be invited to take part in the study.

ELIGIBILITY:
Inclusion Criteria:

- Each participant must meet all of the following inclusion criteria to be enrolled in the study:

1. Male and female patients 18 to 65 years old at screening
2. Must have a diagnosis of MS, and:

   * Patients with RRMS must be on DMT
   * Patients with progressive MS must not be on DMT
3. Participants with RRMS must be on stable DMT (i.e. must not have had a relapse within 1 month prior to the screening visit). Patients on tecfidera, cladribine, ocrelizumab, alemtuzumab, fingolimod or natalizumab must be enrolled with caution, at Chief Investigator's (CI) discretion because of the lymphopenia caused by these drugs and the risk of thrombocytopenia in 1-2 % of people after alemtuzumab
4. OCB positive CSF either from a previous CSF analysis or from the screening CSF analysis
5. Able and willing to give written informed consent and comply with protocol requirements with the understanding that consent may be withdrawn by the patient at any time without prejudice to future medical care.
6. Agree to the use of effective contraception as follows:

   Female patients must:
   * Be postmenopausal for at least 1 year before the screening visit (postmenopausal status confirmed by serum Follicle Stimulating Hormone (FSH) and oestrogen levels at screening or from a historical sample), OR
   * Surgically sterile, OR
   * If they are of childbearing potential, must agree to practice two effective methods of contraception concurrently from the time of signing the informed consent form until 90 days after the last dose of study drug, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence e.g. calendar, ovulation, symptothermal, post-ovulation methods and withdrawal are not acceptable methods of contraception

   Male patients must:
   * Even if surgically sterilized (post-vasectomy with documentation of azoospermia), agree to practice effective barrier contraception during the entire study treatment period and through to 90 days after the last dose of study drug, OR
   * Agree to practice true abstinence when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence e.g. calendar, ovulation, symptothermal, post-ovulation methods and withdrawal are not acceptable methods of contraception
7. Clinical laboratory values:

   1. Absolute neutrophil count (ANC) ≥ 1 x 109/L
   2. Platelet count ≥ 100 x 109/L
   3. Total bilirubin ≤ 1.5 × the upper limit of the normal range (ULN)
   4. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤ 3 × ULN.
   5. Calculated creatinine clearance ≥ 30 mL/min

Exclusion Criteria:

* Participants meeting any of the following exclusion criteria are not to be enrolled in the study:

  1. EDSS > 8.5 at screening
  2. MS relapse within 1 month prior to screening
  3. Female patients who are lactating or have a positive serum pregnancy test at screening
  4. Major surgery within 14 days before baseline
  5. Any clinically relevant malignancy or infection, as per CI/PI (or delegate) decision, including a possible diagnosis of multiple myeloma: raised erythrocyte sedimentation rate (ESR) and positive urine Bence Jones protein at screening
  6. Infection requiring systemic (intravenous) antibiotic therapy or other serious infection within 14 days before study enrolment. Urinary tract infections (UTIs) will be treated prior to baseline and may delay baseline
  7. Evidence of current uncontrolled cardiovascular conditions, including uncontrolled hypertension, uncontrolled cardiac arrhythmias, symptomatic congestive heart failure, unstable angina, or myocardial infarction within 6 months of screening
  8. Systemic treatment, within 14 days before the first dose of ixazomib, with strong Cytochrome P450 Isoform 3A (CYP3A) inducers (rifampin, rifapentine, rifabutin, carbamazepine, phenytoin, phenobarbital), or use of St. John's Wort
  9. History of active hepatitis B or C virus infection, or human immunodeficiency virus (HIV) positive or positive Tuberculin (TB) ELISPOT. If there is positive TB ELISPOT and the TB team decides to treat as latent TB, participants can be reassessed for inclusion after treatment
  10. Any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with the completion of treatment according to this protocol
  11. Known GI disease or GI procedure that could interfere with the oral absorption or tolerance of ixazomib including difficulty swallowing
  12. Diagnosed or treated for malignancy within 2 years before study enrolment or previously diagnosed with another malignancy and have any evidence of residual disease. Patients with non-melanoma skin cancer or carcinoma in situ of any type are not excluded if they have undergone complete resection
  13. Patient has ≥ Grade 3 peripheral neuropathy, or Grade 2 with pain on clinical examination during the screening period
  14. Participation in other clinical trials involving investigational (unlicensed) medicinal products, licensed medicinal products or alternative medicinal therapies, within 30 days of screening and throughout the duration of this trial. Participation in non-interventional, questionnaire or observational studies whilst enrolled in this study is permitted.
  15. Patients that have previously been treated with ixazomib or participated in a study with ixazomib whether treated with ixazomib or placebo
  16. Known allergy to any of the study medications, their analogues, or excipients in the various formulations of any agent
  17. Any pre-existing central nervous system disease or involvement other than MS
  18. History of uncontrolled drug or alcohol abuse within 6 months prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety - Adverse events (AE) will be compared between active and placebo arm | Baseline to 24 months
  1. Proportion of AEs in the Ixazomib versus placebo arm in subjects with Relapsing Remitting Multiple Sclerosis (RRMS)
  2. Proportion of serious AEs (SAEs) in the Ixazomib versus placebo arm in subjects with RRMS
  3. Proportion of AEs in the Ixazomib versus placebo arm in subjects with progressive MS
  4. Proportion of serious AEs (SAEs) in the Ixazomib versus placebo arm in subjects with progressive MS
  5. Proportion of AEs in the Ixazomib versus placebo arm in all subjects (subjects with RRMS and subjects with progressive MS)
  6. Proportion of serious AEs (SAEs) in the Ixazomib versus placebo arm in all subjects (subjects with RRMS and subjects with progressive MS)
Efficacy - the proportion of OCB IgG negative subjects will be compared between active and placebo arm | Baseline to 24 months
  1. Proportion of all subjects (Relapsing Remitting Multiple Sclerosis and progressive Multiple Sclerosis subjects) negative for Oligoclonal Bands Immunoglobulin G (OCB IgG) antibodies measured in Cerebrospinal Fluid (CSF) in the Ixazomib versus placebo arm at 24 months
  2. Proportion of subjects negative for Oligoclonal Bands Immunoglobulin G (OCB IgG) antibodies measured in Cerebrospinal Fluid (CSF) in the Ixazomib versus placebo arm at 24 months in subjects with Relapsing Remitting Multiple Sclerosis (RRMS)
  3. Proportion of subjects negative for Oligoclonal Bands Immunoglobulin G (OCB IgG) antibodies measured in Cerebrospinal Fluid (CSF) in the Ixazomib versus placebo arm at 24 months in subjects with progressive Multiple Sclerosis

SECONDARY OUTCOMES:
Magnetic Resonance Imaging (MRI) | Baseline to 24 months
  Change in T2 lesion load and gadolinium enhancing lesions on brain MRI with Ixazomib versus placebo arm at 24 months
Change In Expanded Disability Status Scale (EDSS) with Ixazomib versus placebo arm at 24 months. The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability. Scoring is based on an examination by a neurologist | Baseline to 24 months
  Change in EDSS with ixazomib versus placebo at 24 months.

OTHER OUTCOMES:
Exploratory endpoint - IgG FLC | Baseline to 24 months
  a. Proportion of all subjects who show reduction in total levels of Immunoglobulin G Free Light Chain (IgG FLC) in Cerebrospinal Fluid (CSF) at 24 months in the Ixazomib versus placebo arm.
Exploratory endpoint - CD19 | Baseline to 24 months
  b. Proportion of all subjects who show change in levels of Cluster of Differentiation antigen 19 (CD 19) at 24 months in the Ixazomib versus placebo arm.
Exploratory endpoint - soluble CD 138 | Baseline to 24 months
  c. Proportion of all subjects who show change in levels of soluble CD 138 at 24 months in the Ixazomib versus placebo arm
Exploratory endpoint - CD 27 | Baseline to 24 months
  d. Proportion of all subjects who show change in levels of soluble CD 27 at 24 months in the Ixazomib versus placebo arm
Exploratory endpoint - neurofilament light chain | Baseline to 24 months
  e. Proportion of all subjects who show change in levels of neurofilament light chain at 24 months in the Ixazomib versus placebo arm
Exploratory endpoint - neurofilament heavy chain | Baseline to 24 months
  f. Proportion of all subjects who show change in levels of neurofilament heavy chain at 24 months in the Ixazomib versus placebo arm
Exploratory endpoint - neopterin | Baseline to 24 months
  g. Proportion of all subjects who show change in levels of neopterin at 24 months in the Ixazomib versus placebo arm
Exploratory endpoint - cytokines profile | Baseline to 24 months
  h. Proportion of all subjects who show change in levels of cytokines profile at 24 months in the Ixazomib versus placebo arm
Exploratory endpoint - GFAP | Baseline to 24 months
  i. Proportion of all subjects who show change in levels of Glial fibrillary acidic protein (GFAP) at 24 months in the Ixazomib versus placebo arm
Exploratory endpoint - NCAM | Baseline to 24 months
  j. Proportion of all subjects who show change in levels of Neural cell adhesion molecule (NCAM) at 24 months in the Ixazomib versus placebo arm
Exploratory endpoint - GAP43 | Baseline to 24 months
  k. Proportion of all subjects who show change in levels of Growth Associated Protein 43 (GAP43) at 24 months in the Ixazomib versus placebo arm
Exploratory endpoint - S100B | Baseline to 24 months
  l. Proportion of all subjects who show change in levels of S100 calcium-binding protein B (S100B) at 24 months in the Ixazomib versus placebo arm

CONTACTS AND LOCATIONS:
Locations (1):
- Royal London Hospital, Barts Health NHS Foundation Trust, London, Greater London, United Kingdom

IPD SHARING:
Plan to Share IPD: No